CLINICAL TRIAL: NCT02165709
Title: Cohort Study of Risk Reducing Salpingectomy (RRS) Versus Standard Tubal Sterilization Among Women Who Desire Sterilization
Brief Title: Cohort Study of Risk Reducing Salpingectomy
Acronym: RRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-0337
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Sterilization, Tubal; Salpingectomy; Ovary; Prevention & Control
MeSH Terms: interventions — Salpingectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Salpingectomy (Experimental): Participants will be offered a risk-reducing salpingectomy, and if they choose this options the surgeon will proceed with a salpingectomy.
  Interventions: Procedure: Salpingectomy
- Traditional sterilization (Active Comparator): Participants will be offered a risk-reducing salpingectomy, and those that choose a traditional sterilization will be in this treatment arm.
  Interventions: Procedure: Traditional sterilization

INTERVENTIONS:
Procedure: Salpingectomy
  Arms: Salpingectomy
Procedure: Traditional sterilization
  Arms: Traditional sterilization

SUMMARY:
Women undergoing surgical sterilization will be interested in risk reducing salpingectomy, and surgeons performing the procedure will be able to successfully complete the salpingectomy.

ELIGIBILITY:
Inclusion Criteria:

* Women > 35 years requesting sterilization as interval procedure OR at time of cesarean delivery
* At least one living child
* English or Spanish speaking
* Sterilization planned as interval (laparoscopic) procedure via Family Planning Clinic services or at time of delivery
* Delivery by cesarean section (planned or following labor)

Exclusion Criteria:

* Age < 30
* Medical complications that increase risk for surgical bleeding (e.g. Idiopathic thrombocytopenic purpura (ITP); von Willebrand disease (vWD); need for prophylactic or therapeutic anticoagulation)

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Percent of women accepting RRS | 12 months
  Determination of patient demand/interest in pursuing RRS for sterilization during 12-month study period

SECONDARY OUTCOMES:
Percent of women with successful RRS completion | 12 months
  Feasibility will be defined as number (%) of successful RRS completion when intended

CONTACTS AND LOCATIONS:
Overall Officials: Matthew L Zerden, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Hosptials, Chapel Hill, North Carolina, United States